

## TRIAL STATISTICAL ANALYSIS PLAN

**Document No.:** 228892 116922 1.0

**BI Trial No.:** 0352-2190

Profiling study for the hepatic cytochrome P450 (CYP) isozymes Title:

CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A in healthy subjects and in patients with stage 4 (F4) liver fibrosis / cirrhosis by the combined administration of the probe substrates (the cocktail) caffeine, warfarin, omeprazole, metoprolol, and

midazolam

(including Protocol Amendment No. 1 [c38905324-02])

**Investigational Product(s):** 

caffeine, warfarin, omeprazole, metoprolol, and midazolam

Responsible trial statistician(s):



Fax:

**Date of statistical** 

09 MAY 2025

analysis plan:

Version: 1.0

Page 1 of 29

#### Proprietary confidential information

© 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 1. TABLE OF CONTENTS

| TITLE PA | AGE1 |
|--------------|--------------------------------------------------|
| 1. | TABLE OF CONTENTS2 |
| LIST OF | TABLES4 |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION8 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY9 |
| 5. | ENDPOINTS |
| 5.1 | PRIMARY ENDPOINTS10 |
| <b>5.2</b> | SECONDARY ENDPOINTS10 |
| 5.2.1 | Key secondary endpoints10 |
| 5.2.2 | Secondary endpoints |
| | v I |
| 5.3.3 | Safety endpoints11 |
| 6. | GENERAL ANALYSIS DEFINITIONS |
| 6.1 | TREATMENTS |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS |
| 6.3 | INTERCURRENT EVENTS |
| 6.4 | SUBJECT SETS ANALYSED15 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS16 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS17 |
| 7. | PLANNED ANALYSIS18 |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS19 |
| <b>7.2</b> | CONCOMITANT DISEASES AND MEDICATION19 |
| 7.3 | TREATMENT COMPLIANCE |
| 7.4 | PRIMARY OBJECTIVE ANALYSIS20 |
| 7.4.1 | Main analysis |
| | CECOND ADVIORUSCIENTE ANALYCIC |
| 7.5 | SECONDARY OBJECTIVE ANALYSIS |
| 7.5.1 | Key secondary objective analysis21 |
| 7.5.2 | Secondary objective analysis21 |
| 7.6.3 | Safety endpoints |
| 7.0.5<br>7.7 | EXTENT OF EXPOSURE22 |
| * · | |


0352-2190

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| 7.8 | SAFETY ANALYSIS | 22 |
|--------------|-----------------------------------------------|----|
| <b>7.8.1</b> | Adverse Events | |
| 7.8.2 | Laboratory data | |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Physical examination | 25 |
| <b>7.9</b> | OTHER ANALYSIS | 25 |
| 7.9.2 | PK analyses | 25 |
| 8. | TIMEPOINT OF RELEASE OF TREATMENT INFORMATION | 26 |
| 9. | REFERENCES | 27 |
| 11. | HISTORY TABLE | 29 |

# **Boehringer Ingelheim**

**Page 4 of 29** 


0352-2190

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# LIST OF TABLES

| Table 6.1: 1 | Analysis phases for statistical analysis of AEs | 13 |
|--------------|--------------------------------------------------|----|
| | Labels defined by study group for tables/figures | |
| | Subject sets analysed | |
| | History table | |

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|---|---|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| ANOVA | Analysis of Variance |
| AST | Aspartate Aminotransferase |
| AUC <sub>0-24</sub> | Area under the concentration-time curve of the analyte in plasma from 0 to 24h |
| AUC <sub>0-96</sub> | Area under the concentration-time curve of the analyte in plasma from 0 to 96h |



BMI Body Mass Index
BP Blood Pressure

CARE Clinical Analysis and Reporting Environment

CIs Confidence Intervals

C<sub>max</sub> Maximum measured concentration of the analyte in plasma

CRF Case Report Form, paper or electronic (sometimes referred to as 'eCRF')

CTCAE Common Terminology Criteria for Adverse Events

CTP Clinical Trial Protocol
CTR Clinical Trial Report

CV Arithmetic Coefficient of Variation

CYP Cytochrome P450

DBLM Database Lock Meeting
DILI Drug induced liver injury

ECG Electrocardiogram


0352-2190

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

| Term | Definition / description |
|--------|----------------------------------------------|
| eDC | Electronic Data Capture |
| EDMS | Electronic Document Management System |
| EMA | European Medicines Agency |
| ES | Enrolled Set |
| FDA | The Food and Drug Administration |
| F/U | Follow-up |
| gCV | Geometric Coefficient of Variation |
| gMean | Geometric Mean |
| ICH | International Conference on Harmonisation |
| INR | International Normalised Ratio |
| iPD | Important protocol devation |
| Max | Maximum |
| Mean | Arithmetic mean |
| MedDRA | Medical Dictionary For Regulatory Activities |
| Min | Minimum |
| N | Number of non-missing observations |
| Nobs | Number of observations |
| P10 | 10 <sup>th</sup> percentile |
| P90 | 90 <sup>th</sup> percentile |
| P-gp | P-glycoprotein I |
| PK | Pharmacokinetics |
| PKS | PK parameter analysis set |
| PR | Pulse rate |
| PT | Preferred Term |
| Q1 | 1 <sup>st</sup> quartile |
| Q3 | 3 <sup>rd</sup> quartile |
| R | Reference |
| RAGe | Report Appendix Generator system |
| REP | Residual Effect Period |
| RNA | Ribonucleic acid |

**RPM** 

Report Planning Meeting


**0352-2190** 228892\_116922\_1.0

| Proprietary confidential inform | ation © 2025 Boehringer Ingelh | eim International GmbH or one | or more of its affiliated companies. |
|---|---|---|---|

| Term | Definition / description |
|--------|--------------------------------------------------|
| SAE | Serious Adverse Event |
| SD | Standard deviation |
| SOC | System Organ Class |
| SOP | Standard Operating Procedure |
| T | Test |
| TMCP | Translational Medicine and Clinical Pharmacology |
| TMF | Trial Master File |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal |
| WHO-DD | World Health Organization Drug Dictionary |

WHO-DD World Health Organization Drug Dictionary

 0352-2190

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 3. INTRODUCTION

Date: 09 MAY 2025, Version 1.0

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This Trial Statistical Analysis Plan (TSAP) assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, and planning of sample size.

Study data as collected in the Case Report Form (eCRF) will be stored in a trial database within the RAVE EDC system. All study data also including external data will then be uploaded to the CDR data warehouse.



 **0352-2190** 

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses as planned in the CTP will be performed and are described in more detail in this TSAP. The following changes compared to the CTP will be made:

According to the study design, the treatment groups incorrectly referred to in the CTP actually correspond to the study groups. Therefore, only the term "study group" is used in the TSAP and the citations from the CTP have been corrected in the TSAP.

Smoking and drinking habits (cf. **CTP Section 5.2.5**) were not captured in the eCRF and will therefore not be reported.

CTP Section 7.2.4.1 incorrectly refers to CTP Section 7.2.3, but should refer to CTP Section 7.2.2 (statistical model):

Further PK endpoints will be analysed descriptively.

The end of the on-treatment phase for reporting adverse events (AEs) was defined based on the residual effect period (REP) specified in **CTP Section 1.2.6** (9 days) and not as erroneously indicated in the **CTP Section 7.2.5** as 10 days.

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

## **Section 2.2 of the CTP:**

Primary endpoint(s) is to determine the following pharmacokinetic parameters for the different components following a single dose of the CYP-cocktail containing caffeine, warfarin, omeprazole, metoprolol, and midazolam.

- $AUC_{0-24}$  (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24 hours) for caffeine, omeprazole, metoprolol, and midazolam
- $AUC_{0-96}$  (area under the concentration time curve of R-warfarin and S-warfarin in plasma over the time interval from 0 to 96 hours)
- $C_{max}$  (maximum measured concentration of the analyte in plasma) for each component of the CYP-cocktail: caffeine, R-warfarin, S-warfarin, omeprazole, metoprolol, and midazolam

## 5.2 SECONDARY ENDPOINTS

## 5.2.1 Key secondary endpoints

This section is not applicable as no key secondary endpoints have been defined in the CTP.

## 5.2.2 Secondary endpoints


This section is not applicable as no secondary endpoints have been defined in the CTP.



 **0352-2190** 

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



## 5.3.3 Safety endpoints

The following safety endpoints have been defined in CTP Section 2.3.2:

- Adverse events (AEs) including clinically relevant findings from the physical examination
- Safety laboratory tests
- 12-lead ECG
- *Vital signs (BP* [blood pressure], *PR* [pulse rate])



 **0352-2190** 

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.



Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENTS

For basic study information on the treatment to be administered and selection of doses, refer to **CTP Section 4**. For information of overall trial design, refer to **CTP Section 3**.

The study is performed as an open-label, single-dose, non-randomised trial. All subjects will receive a single dose of 100 mg caffeine, 5 mg warfarin, 20 mg omeprazole, 50 mg metoprolol, and 2 mg midazolam administered as drug cocktail.

In total, it was planned that 12 healthy subjects and 18 liver cirrhosis patients, of which 12 compensated F4 Child-Pugh A patients and 6 decompensated F4 Child-Pugh B patients, would enter the trial.

### CTP Section 1.2.6:


The Residual Effect Period (REP) of the cocktail is 9 days referring to warfarin, the drug with the longest half-life among the cocktail components.

The following <u>Table 6.1: 1</u> defines the three different phases, screening, on-treatment and follow-up phase, for the statistical analysis of AEs.

Table 6.1: 1 Analysis phases for statistical analysis of AEs

| Study analysis phase | Label | Start (inclusive) | End (exclusive) |
|---|---|---|---|
| Screening <sup>1</sup> | Screening | Date of informed consent | Date/time of administration of study cocktail |
| On-treatment | Cocktail | Date/time of administration of study cocktail | Date/time of<br>administration of<br>study cocktail +<br>residual effect period<br>(9 days)<br>or<br>12:00 a.m. on day<br>after subject's trial<br>termination date,<br>whichever occurs first |
| Follow-up | F/U | Date/time of<br>administration of study<br>cocktail + residual<br>effect period (9 days) | 12:00 a.m. on day<br>after subject's trial<br>termination date |

<sup>&</sup>lt;sup>1</sup> See <u>Section 6.7</u> for definition of baseline, which will be used in the statistical analyses of laboratory data and vital signs.

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

AE summary tables will present results for the on-treatment phase, considering data between start of treatment and end of the REP, as well as AEs starting before cocktail intake and deteriorating under treatment, see **CTP Section 7.2.5**.

In Section 9.4 and Appendix 10.6 (Listings) of the CTR displays, the screening period, as well as the follow-up phase will additionally be included.

Statistical analyses of data such as demography, medical history, concomitant medication, disposition, visit-based data (e.g. vital signs), PK parameters and exploratory biomarkers will be presented by study group.

The labels for the designation of the study groups will be used as displayed in <u>Table 6.1: 2</u>.

Table 6.1: 2 Labels defined by study group for tables/figures

| Study group | | Short label |
|---|---|---|
| 1 | Healthy subjects | Healthy |
| 2 | Compensated F4 Child-Pugh A liver cirrhosis patients | Child-Pugh A |
| 3 | Decompensated F4 Child-Pugh B liver cirrhosis patients | Child-Pugh B |

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

## 6.2 IMPORTANT PROTOCOL DEVIATIONS


Data discrepancies and deviations from the CTP will be identified for all treated subjects. Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the final Report Planning Meeting (RPM). At this meeting, all manual deviations identified at the sites by the Clinical Research Associates and deviations too complex to program will be reviewed by the trial team to decide which are considered important. For definition of important protocol deviations (iPDs), and for the process of identification of these, refer to the BI SOP "Identify and Manage Important Protocol Deviations (iPD)" (2).

The iPD categories are pre-specified in the DV domain sheet. The iPDs will be identified no later than in the RPM, and the iPD categories will be updated as needed. If any iPDs are identified, they are to be summarised into categories and will be captured in the iPD specification file (DV domain) and in the decision log. Both documents will be stored within the Trial Master File in Electronic Document Management System.

0352-2190 Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

The iPDs will be summarised and listed in the CTR.

#### 6.3 INTERCURRENT EVENTS

This section is not applicable as no intercurrent events have been defined in the CTP.

#### 6.4 SUBJECT SETS ANALYSED

The enrolled set (ES), treated set (TS), and pharmacokinetic parameter analysis set (PKS) will be used as defined in CTP Section 7.2:

- Enrolled set (ES): This subject set includes all subjects having signed informed consent and who were screened for inclusion into the study. The enrolled set will be used for analyses of subject disposition.
- *Treated set (TS): The treated set includes all subjects who signed informed consent* and were treated with at least one dose of study drug. The treated set will be used for safety analyses.
- Pharmacokinetic parameter analysis set (PKS): This set includes all subjects in the treated set (TS) who provide at least one PK endpoint that was defined as primary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability (as specified in the following subsection 'Pharmacokinetics'). Descriptive and model-based analyses of PK parameters will be based on the PKS.

The following <u>Table 6.4: 1</u> illustrates the different subject sets used for analyses.

Table 6.4: 1 Subject sets analysed

| | | Subject set | |
|------------------------|--------------|-------------|-----|
| Class of analysis | Enrolled set | Treated set | PKS |
| Pharmacogenomics | | | X |
| Safety endpoints | | X | |
| Disposition | X | | |
| iPDs | | X | |
| Demographic & baseline | | X | |

Details on possible relevant protocol deviations and non-evaluability of plasma concentrations are given in CTP Section 7.2.



228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

The imputation of missing values for safety parameters is not intended. One exception where imputation might be necessary for safety evaluation is AE dates. Missing or incomplete AE dates are imputed according to BI standards (3).

#### CTP Section 7.3.2:

PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.

Missing data and outliers of PK data are handled according to BI standards (4) and (5).

If a subject is removed from or withdraws from the trial prior to the administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF; in addition, trial data will be included in the CRF and will be reported in the CTR.

## Exclusion of PK parameters

The ADS "ADPP" (PK parameters) contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS will include parameters if they are not flagged for exclusion, that is APEXC is equal to "Included".

#### **CTP Section 7.2:**

Exclusion of a subject's data will be documented in the CTR. [...] Plasma concentration data and parameters of a subject which is flagged for exclusion will be reported with its individual values but will not be included in the statistical analyses.

## Exclusion of PK concentrations


The ADS "ADPC" (PK concentrations per time-point or per time-interval) or "ADYC" (PD concentrations per time-point) contains column variables ACEXC and ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to 'ALL CALC', the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to 'DESC STATS' the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition 'TIME VIOLATION' or 'TIME DEVIATION' the value can be used for further analyses based on actual times. If ACEXCO is set to 'HALF LIFE', the value will be excluded from half-life calculation (and, as a consequence, any calculation that relies on  $\lambda z$ ) only; the value is included for all other analyses.

Further details are given in BI-KMED-TMCP-MAN-0014 "Noncompartmental PK/PD Analyses of Clinical Studies" (5) and BI-KMED-TMCP-MAN-0010: "Description of Analytical Transfer Files, PK/PD Data files and ADA files" (6).

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

The last available value determined prior to administration of study cocktail will be defined as baseline.

Adherence to time windows will be checked at the final RPM. Time windows are defined in **CTP Section 6.1**:

The acceptable deviation from the scheduled time for vital signs, ECG, and laboratory tests will be  $\pm$  15 min.

Unscheduled measurements of laboratory data and vital signs data will be assumed to be repeat measurements of the most recent scheduled measurement (e.g. for follow-up or confirmation of a particular value). Therefore, unscheduled measurements will be assigned to the planned time point of the previous scheduled measurement.


**0352-2190** 228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

## 7. PLANNED ANALYSIS

Safety analysis will be performed by the and will be presented in Sections 9.1 to 9.4 of the CTR and in Appendix 10.6 and 10.5.1.

Statistical model-based analysis of PK endpoints will be performed by presented in Section 9.5 of the CTR and in Appendix 10.5.3.

Descriptive data analysis of PK and pharmacogenomics will be performed by the

and will be presented in Section

9.6 and/or 9.7 of the CTR and in Appendix 10.5.5 and/or 10.5.6.

The format of the listings and tables will follow the BI standards ( $\frac{7}{2}$ ) with the exception of those generated for PK-calculations following BI standards for PK/PD analysis ( $\frac{8}{2}$ ).

The individual values of all subjects will be listed, sorted by study group, subject number, and visit. The listings will be included in Appendix 10.6 of the CTR.

For End-Of-Text tables, the set of summary statistics for continuous variables is:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For analyte concentrations and PK parameters, the following descriptive statistics will additionally be calculated:

Nobs number of observations

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

P10 10th percentile
Q1 1st quartile

Q3 3rd quartile


P90 90th percentile

The data format for descriptive statistics of concentrations will be identical to the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Descriptive statistics of PK parameters and biomarker endpoints will be calculated if data from  $N\geq 2$  subjects per study group from at least 1 study group are available.

Statistical model-based analysis will be conducted if data from N≥3 subjects per study group from at least 2 study groups are available.

It should be noted that due to the exploratory nature of the analyses and due to the possibly relatively small number of subjects in a study group, the descriptive statistics or statistical results should be interpreted generally with caution. (When the number of subjects is low, data of single subjects has a higher impact on results.)

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective study group (unless otherwise specified, all subjects in the respective subject set whether they have non-missing values or not).

The precision for percentages should be one decimal point, unless the denominator is smaller than 100 (in all treatment columns), in which case percentages are given in integer numbers. The category missing will be displayed only if there are actually missing values.

Units of variables will be given in the titles or column/row descriptors in brackets (e.g. (mg)).

## 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the report, based on the TS. The data will be summarised by study group and additionally in total for the Appendix 10.5.1.4:1.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases and non-drug therapies will be coded using the latest version of the coding system of the Medical Dictionary for Drug Regulatory Activities (MedDRA). Concomitant medications will be coded using the latest version of the World Health Organization Drug Dictionary (WHO-DD). The coding version number will be displayed as a footnote in the respective output.

Only descriptive statistics are planned for this section of the report, based on the TS. The data will be summarised by study group.

The relevance of the concomitant therapies to the evaluation of PK will be decided no later than at the final RPM.

#### 7.3 TREATMENT COMPLIANCE

#### **CTP Section 4.5:**


Compliance will be assured by administration of trial medication in the study centre under supervision of the investigating physician or a designee by the so-called four-eve principle

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

(two-person rule). For this, one authorised employee of the trial site should witness the administration of trial medication, and – if applicable – its preparation (e.g., reconstitution), if correct dosage cannot be ensured otherwise. The measured plasma concentrations of trial medication will provide additional confirmation of compliance.

Treatment compliance will not be analysed as a specific endpoint. Any deviation from complete intake will be addressed in the final RPM (see <u>Section 6.2</u>) and described in the CTR.

#### 7.4 PRIMARY OBJECTIVE ANALYSIS

Independent of the main objectives stated in the CTP, this section describes further details of the primary endpoint analyses outlined in the CTP.

### 7.4.1 Main analysis

#### Section 7.2.2 of the CTP:

The primary endpoints as specified in section 2.2 will be calculated according to the BI's relevant standards and processes. The analysis will be based on the PKS and will be descriptive in nature.

The statistical model used for the analysis of the primary endpoints will be an analysis of variance (ANOVA) model on the logarithmic scale. That is, the PK endpoints will be log-transformed (natural logarithm) prior to fitting the ANOVA model. This model will include effects accounting for the following sources of variation: '[study] group', age, and BMI. All effect[s] will be considered as fixed. The model is described by the following equation:

$$y_{km} = \mu + \pi_k + age_m + BMI_m + e_{km},$$

where

- $y_{km} = logarithm of response measured on subject m [from study group] k$ ,
- $\mu$  = the overall mean,
- $\pi_k$  = the  $k^{th}$  [study] group effect, i.e. degree of hepatic impairment, k=1 for healthy/normal (Group 1), 2 for Group 2 [Child-Pugh A] or 3 for Group 3 [Child-Pugh B] respectively,,
- $age_m$  = the age of subject m,
- $BMI_m$ = the BMI of the subject m,
- $e_{km}$  = the random error associated with the  $k^{th}$  [study] group effect for subject m
- where  $e_{km} \sim N(0, \sigma_k^2)$  i.i.d,


Point estimates for the ratios of the geometric means (test [T]/reference [R]) for the primary endpoints (see section 2.2) and their two-sided 90 % confidence intervals (CIs) will be provided [where reference is healthy subjects and the test group are the individual patient groups].

For each endpoint, the difference between the expected means for log(T)-log(R) will be estimated by the difference in the corresponding adjusted means (Least Squares Means).

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

Additionally, their two-sided 90% confidence intervals will be calculated based on the residual error from the ANOVA and quantiles from the t-distribution. These quantities will then be backtransformed to the original scale to provide the point estimate and 90 % CIs for each endpoint.

All parameters are calculated and analysed descriptively by study group in addition to the model-based approach.

These analyses will be based on the PKS.



#### 7.5 SECONDARY OBJECTIVE ANALYSIS

## 7.5.1 Key secondary objective analysis

This section is not applicable as no key secondary endpoint has been specified in the protocol.

## 7.5.2 Secondary objective analysis


This section is not applicable as no secondary endpoint has been specified in the protocol.



228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

### 7.6.3 Safety endpoints

Safety endpoints and tolerability will be analysed as described in Section 7.8 of this TSAP.

#### 7.7 EXTENT OF EXPOSURE

Since only a single dose is administered per subject, a listing will be sufficient to give account of the extent of exposure.

### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA at database lock.

The analyses of AEs will be descriptive in nature. For further details on summarisation of AE data, please refer to "Analysis and Presentation of AE data from clinical trials" (9) and "Handling of missing and incomplete AE Dates" (3).

#### **Section 7.2.5 of the CTP:**

Statistical analysis and reporting of adverse events will concentrate on treatment-emergent adverse events, i.e., all adverse events occurring between start of treatment and end of the REP [(9 days)]. Adverse events that start before first drug intake and deteriorate under treatment will also be considered as 'treatment-emergent'.

For details on the treatment definition, see Section 6.1.

According to ICH E3 ( $\underline{10}$ ), in addition to Deaths and serious adverse events, 'other significant' AEs need to be listed in the CTR. These will be any non-serious adverse event that led to an action taken with study drug (e.g. dose reduced or interrupted).

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of adverse events of special interest (AESIs).

The following are considered as AESIs:

## Section 5.2.6.1 of the CTP:

Hepatic injury

Patients with cirrhosis: Hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- Patients with **normal** aminotransferases at baseline:
  - 1. ALT and/or  $AST \ge 3xULN$  combined with a) or b) or c)
    - a) Total bilirubin  $\geq 2xULN$  at the same visit or within 30 days of each other
    - b)  $INR \ge 1.5 \times ULN$  at the same visit or within 30 days of each other
    - c) New-onset or worsening of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, eosinophilia (> 5 %)

OR


228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

- 2. ALT and/or  $AST \ge 5xULN$
- Patients with abnormal ALT, AST, total bilirubin, or INR at baseline:
  - 1. ALT and/or  $AST \ge 2x$  baseline or  $\ge 300$  U/L combined with a) or b) or c)
    - a)  $Total\ bilirubin > 2x\ baseline$
    - b) INR > 1.2x baseline
    - c) New-onset or worsening of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, eosinophilia (> 5 %)

OR

2. ALT and/or  $AST \ge 3x$  baseline

These lab findings constitute a hepatic injury alert. In such instances the testing should be repeated within 48 to 72 hours. If elevations persist, the patients need to be followed up according to the "DILI checklist" provided via eDC. Patients should be followed up until resolution of symptoms or signs in the above stated situations. Patients should also be referred to their hepatologist.

In case of new clinical symptoms of hepatic injury (icterus, unexplained encephalopathy, unexplained coagulopathy, right upper quadrant abdominal pain, etc.) without lab results (ALT, AST, total bilirubin) available, the investigator should make sure these parameters are analysed, if necessary, in an unscheduled blood test. Should the results meet the criteria of hepatic injury alert, the procedures described above should be followed.

For healthy volunteers no AESIs are defined.

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

The intensity (severity) and the causal relationship of AEs are considered according to **CTP Section 5.2.6.1:** 

#### *Intensity (severity) of AEs*

The intensity (severity) of adverse events should be classified and recorded in the CRF according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CTCAE classification ranges from grade 1 to grade 5 (grade 1: mild AE, grade 2: moderate AE, grade 3: severe or medically significant but not immediately life-threatening AE, grade 4: life-threatening AE, grade 5: death related to AE)

#### Causal relationship of AEs


Medical judgement should be used to determine the relationship between the adverse event and the trial treatment, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases, and relevant history.

The frequency of subjects with AEs will be summarised by study group, primary System Organ Class (SOC), and preferred term (PT). Separate tables will be provided for subjects with serious AEs (SAEs), AESIs, drug-related AEs, drug-related SAEs and AE intensity.

The SOCs will be sorted by default alphabetically, PTs will be sorted by frequency (within SOC). The MedDRA version number will be displayed as a footnote in the respective output.

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and PT. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarised.

In addition, frequencies of subjects with non-serious AEs that had an incidence of > 5% for at least one treatment will be summarised by treatment, primary SOC and PT.

## 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and based on BI standards (11).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

#### Section 7.2.5 of the CTP:

Laboratory data will be analysed both quantitatively as well as qualitatively. The latter will be done via comparison of laboratory data to their reference ranges. Values outside the reference range [will be flagged]. [Study] groups will be compared descriptively with regard to distribution parameters as well as with regard to frequency and percentage of patients with abnormal values or clinically relevant abnormal values.

Clinically relevant findings in laboratory data will be reported as baseline conditions (prior to administration of study treatment) or as AEs (after administration of study treatment) if judged clinically relevant by the investigator, and will be analysed as such.

Descriptive statistics of laboratory data including change from baseline (see <u>Section 6.7</u>) will be calculated by planned time point based on the first value of the subject at that planned time point (or assigned to that planned time point). For baseline value, the last measurement before cocktail administration will be used.

## 7.8.3 Vital signs


The analyses of vital signs (BP and PR) will be descriptive in nature.

Clinically relevant findings in vital signs will be reported as baseline conditions (prior to administration of study treatment) or as AEs (after administration of study treatment) if judged clinically relevant by the investigator, and will be analysed as such.

Descriptive statistics of vital signs including change from baseline (see Section 6.7) will be calculated by planned time point based on the first value of the subject at that planned time point (or assigned to that planned time point). For baseline value, the last measurement before cocktail administration will be used.


**0352-2190** 228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

#### **7.8.4** ECG

Clinically relevant findings in ECG will be reported as baseline conditions (prior to administration of study treatment) or as AEs (after administration of study treatment) if judged clinically relevant by the investigator, and will be analysed as such. No separate listing or analysis of ECG data will be prepared.

## 7.8.5 Physical examination

Clinically relevant findings in physical examination will be reported as baseline conditions (prior to administration of study treatment) or as AEs (after administration of study treatment) if judged clinically relevant by the investigator, and will be analysed as such. No separate listing or analysis of physical examination data will be prepared.

#### 7.9 OTHER ANALYSIS



## 7.9.2 PK analyses

The analyte concentrations will be descriptively analysed on the planned sampling times.

## **Section 7.2 of the CTP:**


Only concentration values within the validated concentration range and actual sampling times will be used for the calculation of pharmacokinetic parameters. Concentrations used in the pharmacokinetic calculations will be in the same format provided in the bioanalytical report, (that is, to the same number of decimal places provided in the bioanalytical report).

 **0352-2190** 

228892 116922 1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 8. TIMEPOINT OF RELEASE OF TREATMENT INFORMATION

The treatment information will be loaded into the trial database at trial initiation.

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 9. REFERENCES

| 1. | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2. | <i>BI-VQD-12045_40-413:</i> "Identify and Manage Important Protocol Deviations (iPD)", current version, KMED. |
| 3. | <i>BI-KMED-BDS-HTG-0035:</i> "Handling of Missing and Incomplete AE Dates", current version, KMED. |
| 4. | BI-KMED-TMCP-HTG-0025: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version, KMED |
| 5. | BI-KMED-TMCP-MAN-0014: "Noncompartmental PK/PD Analyses of Clinical Studies", current version, KMED |
| 6. | BI-KMED-TMCP-MAN-0010: "Description of Analytical Transfer Files, PK/PD Data files and ADA files", current version, KMED. |
| 7. | BI-KMED-BDS-HTG-0045: "Standards for Reporting of Clinical Trials and Project Summaries", current version, KMED |
| 8. | BI-KMED-TMCP-OTH-0003: "Graphs and Tables for Clinical Pharmacokinetics and Pharmacodynamic Noncompartmental Analyses", current version, KMED. |
| 9. | <i>BI-KMED-BDS-HTG-0066:</i> "Analysis and Presentation of AE data from clinical trials", current version, KMED. |
| 10. | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version. |
| 11. | BI-KMED-BDS-HTG-0042: "Handling, Display and Analysis of Laboratory Data", current version, KMED. |

 **0352-2190** 

228892 116922 1.0

Proprietary confidential information @ 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.




**0352-2190** 228892\_116922\_1.0

Proprietary confidential information © 2025 Boehringer Ingelheim International GmbH or one or more of its affiliated companies.

# 11. HISTORY TABLE

Table 11: 1 History table

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| 1.0 | 09-MAY-25 | | None | This is the final TSAP. |